CLINICAL TRIAL: NCT05490108
Title: A Two-part, Phase I/II, Randomized, Observer-blinded, Controlled Study to Evaluate the Safety, Reactogenicity, and Immunogenicity of the Recombinant ZR202-CoV and ZR202a-CoV Vaccines Administered at 0 and 28 Days as Compared to Comirnaty ®, and of a Booster Dose of ZR202a-CoV Vaccine in Healthy Adults.
Brief Title: Evaluation of Safety and Immunogenicity of the Recombinant ZR202-CoV and ZR202a-CoV Vaccines in Adults.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zerun Biotechnology Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 202a-COV-2001
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: SARS-CoV-2 Infection; COVID-19
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — ZR202-CoV COVID-19 vaccine; BNT162 Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZR202-CoV - Phase 1 (Experimental): Two doses of SARS-CoV-2 adjuvanted recombinant protein vaccine (prototype), 1 dose each on Day 0 and 28.
  Interventions: Biological: ZR202-CoV
- ZR202a-COV - Phase 1 (Experimental): Two doses of SARS-CoV-2 adjuvanted recombinant protein vaccine (variant), 1 dose each on Day 0 and 28.
  Interventions: Biological: ZR202a-CoV
- Comirnaty® - Phase 1 (Active Comparator): Two doses of Comirnaty® (Pfizer-BioNTech), 1 dose each on Day 0 and 28.
  Interventions: Biological: Comirnaty®

INTERVENTIONS:
Biological: ZR202-CoV — SARS-CoV-2 adjuvanted recombinant protein vaccine (prototype)
  Arms: ZR202-CoV - Phase 1
Biological: ZR202a-CoV — SARS-CoV-2 adjuvanted recombinant protein vaccine (variant)
  Arms: ZR202a-COV - Phase 1
Biological: Comirnaty® — Comirnaty® (Pfizer-BioNTech)
  Arms: Comirnaty® - Phase 1

SUMMARY:
For Phase 1 only. Additional information will be provided when Phase 2 is implemented.

This is a two-part phase I/II, single-center, observer-blind, randomized, controlled vaccine trial to evaluate the safety, reactogenicity, and immunogenicity of the recombinant ZR202-CoV and ZR202a-CoV vaccines administered at 0 and 28 days as compared to Comirnaty®, and of a booster dose of ZR202a-CoV vaccine in healthy adults.

Part 1:

A total of 60 eligible subjects will be randomized in a 1:1:1 ratio into one of the three vaccine groups (ZR202-CoV, ZR202a-CoV, or Comirnaty®), receiving 2 doses vaccination at 28 days interval. To assess safety and preliminary immunogenicity profile after primary series vaccination at pre-defined time points during the study.

The DSMB will review the safety data and provide a recommendation to the Sponsor on whether the safety profile is acceptable for advancing to Part 2.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of both genders, 18 years of age and older, not older than 55 years of age in Part 1.
2. The subject has a BMI (Body Mass Index) ≤30 kg/m2, inclusive, at Screening.
3. Having understood the contents of the ICF and patient information sheet, and having signed the ICF.
4. Free of obvious health problems as established by medical history including physical examination and clinical judgment of the investigator.
5. Clinical laboratory test results within normal reference range, or results with acceptable deviations that are judged to be NCS (Not Clinically Significant) by the investigator. (Part 1 only)
6. Willing to come to study site and/or to receive home visits for the entire study period.
7. Residence in the study area.
8. Female subjects of childbearing potential have used available contraceptive methods during their sexual life within 14 days before enrollment, have no pregnancy plan and will take effective contraceptive measures from enrollment to 1 month after the 2nd vaccination.

Exclusion Criteria:

1. Medical history of COVID-19 or previous vaccination with SARS-CoV-2 vaccine.
2. Fever (body temperature ≥37.5℃/axillary temperature ≥37.3℃) on the day of vaccination or in the 72 hours prior to vaccination.
3. Suffering from any acute clinically significant diseases or being in the acute exacerbation of chronic disease or body temperature ≥37.5℃ (this does not include minor illness such as diarrhea or mild respiratory tract infection) in the 72 hours prior to vaccination.
4. Prior history of allergic reaction or anaphylaxis to any vaccine or drug, e.g., hypersensitivity, urticaria, serious eczema, dyspnea, laryngeal edema, and angioedema etc.
5. Having received or planning to receive any vaccine other than the vaccines used in this clinical study from 28 days prior to the first vaccination to study end (except "vaccines for emergency" such as tetanus vaccine or rabies vaccine).
6. Having participated in or planned to participate in clinical studies of other drugs from 28 days prior to the 1st vaccination to study end (6 months after the 2nd vaccination in Part 1).
7. Presence of uncontrolled chronic pulmonary, cardiovascular, renal, hepatic, neurologic, hematologic, or metabolic (including diabetes mellitus) disorders, which would include the potential subject in a high-risk category for SARS-CoV-2 infection and/or its complications as judged by the investigator.
8. Having hereditary hemorrhagic tendency or coagulation dysfunction (e.g., cytokine defects, coagulation disorders or platelet disorders), or history of significant bleeding, or history of intramuscular injection or venipuncture injury.
9. Known medical history or a previous diagnosis of thrombosis including thrombocytopenia.
10. Known medical history or diagnosis confirming that subjects have diseases affecting immune system function, including cancer (except skin basal cell carcinoma), congenital or acquired immunodeficiency (e.g., infection with HIV [Human Immunodeficiency Virus]), uncontrolled autoimmune disease.
11. Asplenia or functional asplenia.
12. Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying agents within 90 days prior to the administration of study vaccines (including systemic corticosteroids, this means prednisone, or equivalent, ≥0.5 mg/kg/day; topical steroids including inhaled steroids are allowed).
13. Having received immunoglobulins and/or blood products within 3 months prior to the 1st vaccination in this study.
14. Planning to permanently move from the local area before study completion or leave the local area for a long time during the period of study visits.
15. Positive for the pregnancy test (a pregnancy test will be required before each vaccination for all women of childbearing potential) or lactation.
16. Previous inclusion of 5 family members in the study (i.e., subjects belonging to the same family - biological father, mother, child, and brothers and sisters may be included up to a maximum of 5 members from the same family).
17. Any chronic disease, condition, or criteria that in the opinion of the investigator might compromise the wellbeing of the subject or the compliance with study procedures or interfere with the outcome of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-06-02 (Actual); Primary Completion 2022-09-26 (Actual); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects reporting solicited AEs within 7 days after each vaccination (Part 1) | 7 days after the first or second vaccination
Percentage of subjects reporting unsolicited AEs within 28 days after each vaccination (Part 1) | 28 days after the first or second vaccination
Occurrence of out-of-normal range clinical laboratory test results (including change from baseline values) 14 days post vaccination - (Part 1) | Screening Visit, 14 days after the 1st and 2nd vaccinations at Day 14 and Day 42, and 28 days after both vaccinations at Day 28 and Day 56

SECONDARY OUTCOMES:
Immunogenicity as assess for SARS-CoV-2 specific neutralizing antibodies titers 28 days after each vaccination as measured by neutralization assay | Day 28 and Day 56
Percentages of subjects reporting SAEs, AESIs (including COVID-19), MAAEs | From 1st vaccination until 6 months after the 2nd vaccination (Part 1)
Immunogenicity as assess for SARS-CoV-2-specific anti-S protein IgG binding antibodies 28 days after each vaccination as measured by ELISA. | Day 28 and Day 56

CONTACTS AND LOCATIONS:
Overall Officials: Samba Sow, Principal Investigator — Center for Vaccine Development - Mali
Locations (1):
- Center for Vaccine Development-Mali, Bamako, Mali